CLINICAL TRIAL: NCT06790667
Title: Comparative Effectiveness of Low Level Laser Therapy and Transcutaneous Electrical Nerve Stimulation on Pain and Mouth Opening in Temporomandibular Disorders Based Upon Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
Brief Title: Comparison of Low-Level Laser Therapy and Transcutaneous Electrical Nerve Stimulation for Myofascial Pain in Temporomandibular Disorders
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, ARHUM BUTT, Postgraduate Resident, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIVERSITY OF HEALTH SCIENCES
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Temporomandibular Disorders
Keywords: Randomized clinical trial; temporomandibular disorder; myofascial pain; Low-level laser therapy; Transcutaneous Electrical Nerve Stimulation; Jaw Pain Treatment; Mouth opening improvement
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants shall be randomly assigned to receive either:
  Low-Level Laser Therapy (LLLT), or Transcutaneous Electrical Nerve Stimulation (TENS).
  Both groups will be monitored for outcomes like pain reduction and mouth opening improvement over the same timeline, with no participant switching between treatments.
  This approach ensures unbiased comparison of the effectiveness of LLLT and TENS in treating myofascial pain in Temporomandibular Disorders (TMD).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Other): Participants in this arm will receive LLLT for the treatment of myofascial pain associated with TMD.
  Interventions: Device: Low Level Laser Therapy
- Group B (Experimental): Participants in this arm will receive TENS for the treatment of myofascial pain associated with TMD.
  Interventions: Device: Transcutaneous Pulsed Electrical Stimulation (Device: Nu Eyne M02)

INTERVENTIONS:
Device: Low Level Laser Therapy — Participants in this arm will receive Low-Level Laser Therapy (LLLT) using a Gallium Aluminum Arsenide (GaAlAs) semiconductor diode laser. The treatment involves a wavelength range of 650-808 nm with a power output of 775 mW. The therapy is administered by exposing tender points around the temporomandibular joint (TMJ) to the laser for 2 minutes per session. Each participant will receive treatment on alternate days (three sessions per week) over the course of three weeks. The goal is to assess the effectiveness of LLLT in reducing pain and improving mouth opening in patients with myofascial pain associated with Temporomandibular Disorders (TMD).
  Arms: Group A
Device: Transcutaneous Pulsed Electrical Stimulation (Device: Nu Eyne M02) — Participants in this arm will undergo Transcutaneous Electrical Nerve Stimulation (TENS), utilizing a four-electrode unit. The device will be set to deliver electrical impulses at a frequency of 150 Hz with a pulse width of 200 µs. Electrodes will be placed over the cutaneous region between the TMJ and coronoid process to stimulate the trigeminal and facial nerves. Each treatment session will last 15 minutes and occur on alternate days, three times a week for three weeks. This therapy aims to provide pain relief and improve jaw function for patients suffering from myofascial pain associated with TMD.
  Arms: Group B

SUMMARY:
Myofascial pain is the most common form of temporomandibular disorder (TMD) encountered in maxillofacial practice. Treatment options range from conservative management to open surgical procedures, with physical therapies identified as the safest and most effective. Among these, transcutaneous electrical nerve stimulation (TENS) is a widely used technique, while low-level laser therapy (LLLT) is a recent therapeutic advancement. This study is designed to compare the efficacy of these two therapies, aiming to identify the more effective option.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted at the Oral and Maxillofacial Surgery department, Punjab Dental Hospital, Lahore. Sample size of 40 patients will be selected through convenience sampling and divided into two equal groups, based on computergenerated random numbers. A written consent will be obtained from all the participants. Group A will receive LLLT, while Group B will receive TENS. The primary variables like pain score and mouth opening will be recorded preoperatively and during followup sessions. The proforma used for data collection will be designed, tailored to the needs of this study based on standard Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). Both groups will receive their assigned therapies on alternate days for three weeks, with evaluations at 1st, 3rd, and 4th weeks post-treatment. All collected data will be entered into SPSS version 25 for statistical analysis. Independent sample t-test will be used to compare the mean pain score and mouth opening between the two groups. Repeated measures ANOVA will be applied to compare the primary variables in both groups on all follow-ups. P-value ≤0.05 will be considered as significant.

This study aims to offer tailored insights and practical recommendations, potentially improving patient care by providing safer and non-invasive alternatives to more invasive procedures thus enhancing overall treatment strategies. It is assumed that expected results shall be in favor of the LLLT group. Possible limitations may include failure of patients to come for multiple sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed cases of myofascial pain in TMD patients, which fall under diagnostic criteria (DC/TMD).
2. Myofascial pain that persists for more than 3 months.
3. Involvement of trigger points in the masseter and temporalis muscles.
4. Impaired or limited mouth opening (less than 35mm).

Exclusion Criteria:

1. Congenital abnormality or neoplastic condition around TMJ.
2. Recent history of trauma affecting head and neck region.
3. Patients with known dermatological disorders (eczema, psoriasis).
4. Patients with pacemakers and cardiovascular diseases.
5. Epileptic patients.
6. Patients allergic to adhesive tapes or electrodes of TENS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (VAS Score) | 6 months
  Change in pain intensity as measured by the Visual Analog Scale (VAS), a 10 cm scale ranging from 0 (no pain) to 10 (worst possible pain) Unit of Measure: Centimeters (cm) Time Points: Pre-treatment, 1st week, 3rd week, and 4th week.
Mouth Opening (Active Interincisal Distance) | 6 months
  Change in active interincisal distance, measured using a ruler from the upper to lower incisal edges during maximum unassisted mouth opening.
  Unit of Measure: Millimeters (mm). Time Points: Pre-treatment, 1st week, 3rd week, and 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Arhum Butt, Bachelor of Dental Surgery, Principal Investigator — University of Health Sciences Lahore

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share IPD because of ethical considerations, limited resources for data preparation, and potential risks of data misuse or misinterpretation.